CLINICAL TRIAL: NCT06863467
Title: A Phase 1b, Randomized, Placebo-Controlled, Single-Blind, Single Ascending Dose Study in Subjects With Stage 3 or 4 Chronic Kidney Disease
Brief Title: Evaluation of the Safety and Tolerability of Gemini in Subjects With Stage 3-4 Chronic Kidney Disease.
Acronym: PRIME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Revelation Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RVL-CKD01
Record Dates: First submitted 2025-02-21; First posted 2025-03-07 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Renal Insufficiency, Chronic; Chronic Kidney Disease stage3; Chronic Kidney Disease stage4
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low dose of intravenous Gemini infused once over 10-15 minutes. (Experimental): Cohort 1, 8 subjects (6 active, 2 placebo)
  Interventions: Drug: Intravenous Gemini; Drug: Intravenous placebo
- Mid-level dose of intravenous Gemini infused once over 10-15 minutes. (Experimental): Cohort 1, 8 subjects (6 active, 2 placebo)
  Interventions: Drug: Intravenous Gemini; Drug: Intravenous placebo
- High dose of intravenous Gemini infused once over 10-15 minutes. (Experimental): Cohort 1, 8 subjects (6 active, 2 placebo)
  Interventions: Drug: Intravenous Gemini; Drug: Intravenous placebo
- Optional High dose of intravenous Gemini infused once over 10-15 minutes. (Experimental): Cohort 1, 8 subjects (6 active, 2 placebo)
  Interventions: Drug: Intravenous Gemini; Drug: Intravenous placebo

INTERVENTIONS:
Drug: Intravenous Gemini — Single ascending intravenous dose infused once over 10-15 minutes.
  Other Names: Phosphorylated hexaacylated disaccharide; PHAD
Drug: Intravenous placebo — Intravenous sugar solution infused in a single dose over 10-15 minutes.
  Other Names: D5W

SUMMARY:
Gemini is being evaluated in a placebo controlled, single dose, escalating dose study to evaluate the safety and tolerability of intravenous Gemini in adult subjects with stage 3 or 4 chronic kidney disease. Pharmacokinetics will be evaluated and measurements of the effect of Gemini on pharmacodynamic activity will be measured to assess changes in potential pharmacodynamic markers.

DETAILED DESCRIPTION:
Design: Randomized, Placebo Controlled, Single Blind, Single-Ascending Dose Study in Patients with Stage 3-4 CKD.

This study is planned as a placebo controlled, single dose, escalating dose study to evaluate the safety and tolerability of intravenous Gemini in adult subjects with stage 3 or 4 chronic kidney disease. This study will enroll up to 40 subjects in up to 5 cohorts. Each cohort will consist of 8 unique subjects, 6 assigned to Gemini and 2 assigned to placebo. All subjects will provide written informed consent and be screened for eligibility before enrollment. All eligibility criteria must be met prior to dosing.

On Day 1, each study subject will receive a single IV dose (each total dose volume = 20 mL) via syringe pump for at least 10 minutes but not longer than 15 minutes and as per the institution's standard method. Time 0 starts once the entire dose is administered and the line has been flushed to ensure any residual drug is delivered.

A Safety Review Committee (SRC) will assess safety and tolerability including AEs, after at least 6 subjects in each cohort have completed Day 8 to determine the subsequent cohort dose. If a grade 3 or higher adverse event is not experienced, as determined by the SRC, or the criteria for stopping dosing has not been met at a given cohort dose level, dose escalation will proceed to the next cohort and dose level.

Dosing will continue until any cohort experiences a dose limiting toxicity (DLT), defined as a dose that causes any grade 3 or higher adverse event, or stopping criteria is met or the highest dose as determined in the Phase 1 study has been tolerated. If a dose is stopped due to a DLT or stopping criteria, cohorts scheduled at a higher dose will not be utilized. The SRC will meet to review safety and tolerability data and may determine if a lower dose can be given. This dose will be documented in the minutes and a dose recommendation memo which will be provided to the clinical sites.

Once the maximum tolerated dose is determined, the dose will be repeated (Cohort 4) for a total of 16 subjects dosed at the highest level tolerated. The repeated dose cohort will consist of 8 unique subjects, 6 assigned to Gemini and 2 assigned to placebo. If the maximum tolerated dose is reached within the first 2 cohorts, the dose will be repeated until a minimum of 32 subjects are enrolled.

If the highest dose determined in the Phase 1 study is tolerated, optional higher dosing of may be administered as determined by the SRC, or the same dose will be repeated.

All visits will be conducted as an outpatient or via telephone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 to ≤ 80 years of age at screening
* Willing and able to provide written informed consent
* eGFR of ≥ 15 and ≤ 60 per
* Female subjects must be of non-childbearing potential or using a medically acceptable contraceptive regimen
* Male subjects must be surgically sterile or using a medically acceptable contraceptive regimen
* Willing and able to tolerate IV infusions and multiple blood draws
* Willing to comply with the study schedule, restrictions, and requirements

Exclusion Criteria:

* CKD Secondary to or associated with any of the following:

  1. History of rapidly progressive glomerulonephritis (RPGN)
  2. Glomerulonephritis requiring any use of immunosuppression in the last 6 months
* Body mass index ≤ 19.0 kg/m2 or ≥ 40.0 kg/m2
* Currently taking a sodium/glucose cotransporter-2 inhibitor (SGLT2i) or non-steroidal mineralocorticoidantagonist (MRA) requiring dose adjustments within 12 weeks prior to Day 1 or if dose is anticipated to change
* Currently taking tumor necrosis factor (TNF) inhibitors, TNF blocker, interleukin-6 (IL-6) blockers or interleukin-1 (IL-1) blocking drugs
* Receiving steroids or any other immunosuppressive agent or anti-inflammatory drugs
* Currently taking an angiotensin-converting enzyme inhibitor (ACEi) and/or an angiotensin II receptor blocker (ARB) requiring dose adjustments
* Any use of direct renin inhibitors;
* Live vaccinations within 3 months prior to the start of the trial or expected during the trial
* Received a mRNA vaccine within 4 weeks
* Uncontrolled diabetes (HbA1c > 11.0%)
* Clinical laboratory results of ALT and/or AST that are > 2.5X upper limit of normal (ULN)
* Clinical Laboratory results of Total bilirubin that is > 1.5X the ULN
* Has a Urine Albumin-to-Creatinine Ratio (uACR) level > 3000 mg/g
* Age-related macular degeneration (AMD), diabetic macular edema or active diabetic proliferative retinopathy that was likely to require treatment during the trial
* Uncontrolled hypertension
* New York Heart Association Class IV congestive heart failure
* Any organ transplant recipient, or a planned transplant during the study
* Currently has known Hepatitis B or uncontrolled human immunodeficiency virus (HIV) or uncontrolled Hepatitis C virus (HCV) that may interfere with the study
* Myocardial infarction, acute coronary syndrome, or stroke within 6 months
* History of myelodysplastic syndrome
* History of deep vein thrombosis (DVT) that required active treatment in the last 6 months. Superficial thrombosis is not excluded
* History of hemosiderosis or hemochromatosis
* History of rheumatoid arthritis or systemic lupus erythematosus (SLE)
* History of drug use that may interfere with the study or study result
* Red cell transfusion within 12 weeks
* History of malignancy in the previous 5 years except for curatively resected basal cell carcinoma of skin, squamous cell carcinoma of skin or cervical carcinoma in situ
* Coronavirus disease 2019 (COVID-19) diagnosis within 1 month
* Evidence of active infection unless subject is appropriate for this study per the Investigator
* Life expectancy less than 6 months
* Intolerance to study medication
* Pregnancy or lactation
* Received treatment with any investigational product in any clinical study within 30 days prior to administration of study drug or five half-lives, whichever is longer
* In the opinion of the Investigator or identified Sub-I(s), any other disease processes or confounding variables that would inappropriately alter the outcome of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Effect of Gemini versus placebo on the incidence of treatment-emergent adverse events. | From time of dose to Day 8
  Collection of side effects reported by subjects.
Effect of Gemini vs placebo on electrical activity of the heart. | From time of dose to Day 8
  Safety measure for change in the electrical activity of the heart over a period of time using electrodes placed on the skin and recorded by electrocardiogram (ECG) after resting for at least 10 minutes in a quiet setting without distractions in a semi-supine position.
Effect of Gemini versus placebo on blood pressure. | From time of dose to Day 8
  Safety measure for change in blood pressure after 5 minutes of rest in a supine, semi-supine or sitting position.
Number of participants with abnormal laboratory hematology test results. | From time of dose to Day 8
  Clinically significant changes in blood hematology levels.
Number of participants with abnormal laboratory chemistry tests results. | From time of dose to Day 8
  Clinically significant changes in blood chemistry levels.
Number of participants with abnormal laboratory urine tests results. | From time of dose to Day 8
  Clinically significant changes in urine.
Effect of Gemini versus placebo on inflammation in the body. | From time of dose to Day 8
  Measurement of erythrocyte sedimentation rate in the blood.
Effect of Gemini versus placebo on inflammation. | From time of dose to Day 8
  Measurement of N-terminal pro b-type natriuretic peptide in the blood.
Effect of Gemini versus placebo on the inflammatory state of CKD subjects. | From time of dose to Day 8
  Measurement of highly sensitive C-reactive Protein in the blood.
Effect of Gemini versus placebo on kidney damage. | From time of dose to Day 8
  Measurement of urine albumin creatinine ratio.
Effect of Gemini versus placebo on heart rate. | From time of dose to Day 8
  Safety measure for change in heart rate (bpm) after 5 minutes of rest in a supine, semi-supine or sitting position.
Effect of Gemini versus placebo on body temperature. | From time of dose to Day 8
  Safety measure for change in body temperature (Celsius) after 5 minutes of rest in a supine, semi-supine or sitting position.
Effect of Gemini versus placebo on respiration. | From time of dose to Day 8
  Safety measure for change in respiration rate after 5 minutes of rest in a supine, semi-supine or sitting position.
Number of participants with abnormal physical exam findings. | From time of dose to Day 8
  Clinically significance changes in general appearance.
Number of participants with abnormal mental physical exam findings. | From time of dose to Day 8
  Clinically significant changes in mental status.
Number of participants with abnormal physical exam findings above the shoulders. | From time of dose to Day 8
  Clinically significant changes with HEENT (head, eyes, ears, nose, throat).
Number of participants with abnormal physical exam findings of the skin. | From time of dose to Day 8
  Clinically significant changes in the dermatologic system.
Number of participants with abnormal physical exam findings of the heart. | From time of dose to Day 8
  Clinically significant changes in the cardiovascular system.
Number of participants with abnormal physical exam findings of the lungs. | From time of dose to Day 8
  Clinically significant changes in the respiratory system.
Number of participants with abnormal physical exam findings of the digestive system. | From time of dose to Day 8
  Clinically significant changes in the gastrointestinal system.
Number of participants with abnormal physical exam findings of the body's support structure. | From time of dose to Day 8
  Clinically significant changes in the musculoskeletal system.
Number of participants with abnormal physical exam findings of the nervous system. | From time of dose to Day 8
  Clinically significant changes in the neurological system.

SECONDARY OUTCOMES:
Peak observed concentration of Gemini. | From time of dose to Day 8
  Measurement of maximum observed concentration (Cmax) in blood over intervals of time.
Time for Gemini to reach to maximum observed concentration. | From time of dose to Day 8
  Measurement of time to maximum observed concentration (Tmax) over intervals of time.
Total amount of Gemini that enters the systemic circulation after administration. | From time of dose to Day 8
  Measurement of area under the concentration-time curve (AUC0-t) over intervals of time.
Total Gemini exposure across time. | From time of dose to Day 8
  Measurement of area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) over intervals of time.
The amount of time required for the plasma concentration of Gemini to decline by 50% . | From time of dose to Day 8
  Measurement if apparent terminal elimination half-life (t1/2) over intervals of time.
Volume of Gemini required to be uniformly distributed throughout the body. | From time of dose to Day 8
  Measurement of blood volume of distribution (Vd) over intervals of time.
Rate which Gemini is removed from the human system. | From time of dose to Day 8
  Measurement of elimination rate constant (Kel) over intervals of time.

OTHER OUTCOMES:
Effect of Gemini versus placebo on serum biomarkers for traditional assessment of inflammation. | From time of dose to Day 8
  Measurements of hsCRP, IL-1 beta, IL-6 and TNF-alpha in blood over time.
Effect of Gemini versus placebo on serum biomarkers that measure activity. | From time of dose to Day 8
  Measurement of NGAL and IL-1 receptor antagonist in the blood over time.
Effect of Gemini versus placebo on urine biomarkers. | From time of dose to Day 8
  Measurement, if necessary, of hsCRP, IL-1 beta, IL-6, and TNF-alpha, NGAL and IL-1 receptor antagonist as dictated by serum biomarker measurement results.
Assessment of Gemini versus placebo on attenuation of inflammatory response. | Day 1 to Day 2.
  Measurement of peripheral blood mononuclear cells response ex vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Executive Officer, Study Director — Revelation Biosciences, Inc
Locations (3):
- United States (3):
  - California Institute of Renal Research, Chula Vista, California
  - California Institute of Renal Research, La Mesa, California
  - Clinical Advance Center, PLLC, San Antonio, Texas